CLINICAL TRIAL: NCT06445244
Title: The Effects of α-ketoglutarate on Blood Pressure and Endothelial Function in Hypertensive Patients
Brief Title: α-ketoglutarate in Patients With Hypertension
Acronym: AKGHTN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Tao (Other)
Responsible Party: Sponsor-Investigator, Jun Tao, Guangxi Hospital Division of The First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-IIT-2024-001
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- α-KG group (Experimental): AKG Double Wood® + lifestyle modification
  Interventions: Dietary Supplement: Alpha-ketoglutarate supplied as 1000mg capsule; Behavioral: Behavioral: Lifestyle modification
- Control group (Other): Lifestyle modification only
  Interventions: Behavioral: Behavioral: Lifestyle modification

INTERVENTIONS:
Dietary Supplement: Alpha-ketoglutarate supplied as 1000mg capsule — AKG Double Wood® + lifestyle modification AKG Double Wood®: 500mg, qd, for one months. Lifestyle modification: intake 1400-1600 kcal/day: 54% carbohydrates, 24% proteins, 22% lipids, 108 mg cholesterol, 35 g fiber; avoid smoking and alcohol consumption; performing aerobic activity 4 days per week such as 45 min on a stationary bicycle.
  Arms: α-KG group
Behavioral: Behavioral: Lifestyle modification — Lifestyle modification: intake 1400-1600 kcal/day: 54% carbohydrates, 24% proteins, 22% lipids, 108 mg cholesterol, 35 g fiber; avoid smoking and alcohol consumption; performing aerobic activity 4 days per week such as 45 min on a stationary bicycle.

SUMMARY:
Cardiovascular and cerebrovascular diseases are most terrible killers endangering the health of Chinese residents, and hypertension is the most important risk factor. Hypertension related microvascular rarefaction and endothelial dysfunction are the common pathological basis and initiation of cardiovascular and cerebrovascular disease. Therefore, reducing blood pressure and delaying or reversing endothelial dysfunction is an effective way to treat hypertension and prevent cardiovascular disease. Alpha-ketoglutarate (αKG) is a critical metabolic intermediate in the tricarboxylic acid (TCA) cycle, involves in diverse cellular biological activities, such as central metabolism, antioxidative defense, epigenetic regulation, and cell proliferation. The latest research found that with the growth of age, the level of αKG is decreasing, and increasing the content of αKG can prolong the life of multiple species including human. Recent clinical trials found that αKG supplementation can effectively improve the level of αKG in cells, delay aging, improve the metabolic process of cells without adverse reactions. However, the effect of αKG supplementation on reducing blood pressure and protecting vascular endothelial function has not been reported. Therefore, this study aims to focus on hypertension, a major chronic disease, and to observe the effects of αKG supplementation on endothelial function and blood pressure in patients with hypertension, so as to provide a new treatment strategy for hypertension and associated endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1、 Primary hypertension (office blood pressure: systolic blood pressure 130～159 mmHg and/or diastolic blood pressure 80～99 mmHg, which meets the diagnostic criteria of hypertension class 1 of 2018AHA hypertension guidelines) and accompanied by vascular dysfunction (FMD<5%); 2、 Age between 18 and 65 years old; 3, Not using any drugs and dietary supplements that affect blood pressure and vascular endothelial function in the last 3 months, mainly including antihypertensive, lipid-lowering, hypoglycemic drugs and natural plant extract antioxidants; 4、 Voluntarily sign the informed consent form after fully understanding the purpose and process of the study, disease characteristics, drug effects, methods of relevant examinations, and potential risks/benefits of the study.

Exclusion Criteria:

1. Presence of secondary hypertension (those who have been diagnosed with secondary hypertension in the past and have not been definitively cured, and if secondary hypertension is suspected, a complete examination is required to exclude common secondary hypertension, including renal hypertension (renal parenchymal lesions, renal artery stenosis), primary aldosteronism, Cushing's syndrome, pheochromocytoma, aortic constriction, and severe obstructive sleep apnea);
2. Acute myocardial infarction within the past 6 months;
3. recent history of stroke (within 6 months); 4, Dilated heart disease, hypertrophic cardiomyopathy, rheumatic heart disease, congenital heart disease, severe heart valve disease (severe valve stenosis and or regurgitation);

5. patients with a combination of serious physical illnesses, such as cancer; 6, Severe hepatic or renal dysfunction (ALT and or AST) ≥ 3 times the upper limit of normal, or dialysis end-stage renal disease or eGFR < 30 ml/min/1.73 m2, or serum creatinine > 2.5 mg/dL [> 221 μmol/L]); 7. Symptomatic heart failure or reduced left ventricular ejection fraction (<40%) within the past 6 months; 8. History of hypersensitivity to the study drug or to its components after administration; 9. Participating in other clinical studies; 10. Patients with mental illness who are unable to cooperate; 11, Pregnant, lactating or expectant mothers;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Effect of αKG on flow mediated dilation （FMD） | Up to 1 month
  Change of FMD between αKG-treated participants and non-αKG-treated participants
Effect of αKG on brachial-ankle pulse wave velocity （baPWV） | Up to 1 month
  Change of baPWV between αKG-treated participants and non-αKG-treated participants

SECONDARY OUTCOMES:
Effect of αKG on blood pressure | Up to 1 month
  Change of systolic blood pressure and diastolic blood pressure between αKG-treated participants and non-αKG-treated participants
Effect of αKG on serum αKG levels | Up to 1 month
  Change of serum αKG levels between αKG-treated participants and non-αKG-treated participants
Effect of αKG on retinal vascular density | Up to 1 month
  Change of retinal vascular density between αKG-treated participants and non-αKG-treated participants

CONTACTS AND LOCATIONS:
Overall Officials: Xia Wenhao, MD, PhD, Study Chair — Guangxi Hospital Division of The First Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Wenhao Xia, Guangxi, Nanning, China

IPD SHARING:
Plan to Share IPD: No